CLINICAL TRIAL: NCT02500212
Title: OPEN-LABEL, MULTICENTRE, RANDOMIZED CLINICAL TRIAL TO COMPARE THE PHARMACOKINETICS OF ENVARSUS® TABLETS AND ADVAGRAF® CAPSULES ADMINISTERED ONCE DAILY IN ADULT DE-NOVO KIDNEY TRANSPLANT PATIENTS
Brief Title: Pharmacokinetic Study of ENVARSUS in Adult De-novo Kidney Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCD-06235AA1-02; 2014-005572-28 (EudraCT Number)
Record Dates: First submitted 2015-07-07; First posted 2015-07-16 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Organ or Tissue Transplant; Complications
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ENVARSUS tablets (Experimental): Envarsus® (tacrolimus) prolonged-release tablets provided in 0.75 mg, 1.0 mg and 4.0 mg dose strengths.
  Envarsus® tablets will be administered orally once daily in the morning
  Interventions: Drug: ENVARSUS®
- ADVAGRAF capsules (Active Comparator): Advagraf® (tacrolimus) prolonged-release hard capsules provided in 0.5 mg, 1.0 mg, 3.0 mg and 5.0 mg dose strengths.
  Advagraf® capsules will be administered orally once daily in the morning
  Interventions: Drug: ADVAGRAF®

INTERVENTIONS:
Drug: ENVARSUS®
  Arms: ENVARSUS tablets
Drug: ADVAGRAF®
  Arms: ADVAGRAF capsules

SUMMARY:
Open-label, multicentre, randomized clinical trial to compare the pharmacokinetics of ENVARSUS® tablets and ADVAGRAF® capsules administered once daily in adult de-novo kidney transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of a kidney transplant from a deceased donor or a living donor

Exclusion Criteria:

* Recipient of any transplanted organ other than a kidney;
* Recipients of a bone marrow or stem cell transplant;
* Recipients of a kidney from a cardiac death donor;
* Recipients of a kidney from an ABO incompatible donor;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Tacrolimus Area under the curve (AUC 0-24h)r h*pg/mL | pre-dose, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 20.0, 24.0 hr post-dose

SECONDARY OUTCOMES:
Tacrolimus concentration 24 hours post-dose (C24hr) pg/mL | 24.0 hr post-dose
  Whole blood trough drug concentration 24hour post dose
Serum creatinine (mg/dL) | before dosing
estimated glomerular filtration rate (eGFR) mL/min; | before dosing
Heart Rate, (beats per minute) | before dosing
Qt (milliseconds) | before dosing

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Nephrology Department Hopital La Cavale Blanche, Brest
  - Clinique de Nephrologie CHU Grenoble, Grenoble
  - CHU Limoges, Limoges
  - Service de Nephrologie, Montpellier
  - Unité de transplantation rénale -Hopital Pasteur, Nice
  - Nephrology department CHU de Saint-Etienne Hospital Nord, Saint-Etienne
  - CHU Rangueil, 1 avenue J Poulhes TSA 50032., Toulouse

REFERENCES:
- [Result] Kamar N, Cassuto E, Piotti G, Govoni M, Ciurlia G, Geraci S, Poli G, Nicolini G, Mariat C, Essig M, Malvezzi P, Le Meur Y, Garrigue V, Del Bello A, Rostaing L. Pharmacokinetics of Prolonged-Release Once-Daily Formulations of Tacrolimus in De Novo Kidney Transplant Recipients: A Randomized, Parallel-Group, Open-Label, Multicenter Study. Adv Ther. 2019 Feb;36(2):462-477. doi: 10.1007/s12325-018-0855-1. Epub 2018 Dec 14. PMID 30552587
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2014-005572-28